CLINICAL TRIAL: NCT03958292
Title: Evaluation of Conjunctival Flora Alteration in Patients Undergoing Cataract Surgery
Brief Title: Conjunctival Flora Before Cataract Surgery: a Microbiological Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Sacra Famiglia - Fatebenefratelli Erba (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OSFFE_OCU_IO18
Record Dates: First submitted 2019-05-08; First posted 2019-05-22 (Actual); Last update posted 2019-05-22 (Actual); Status verified 2019-05

CONDITIONS: Endophthalmitis Following Cataract Surgery
Keywords: Cataract; Endophthalmitis; Microbiological evaluation
MeSH Terms: conditions — Cataract; Endophthalmitis

STUDY DESIGN:
Intervention Model Description: Each patient has self-control of the IODIM treatment in the eye undergoing to cataract surgery with the contralateral eye. Microbiological studies will be performed by means of conjunctival swabs evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients undergoing routine cataract surgery (Experimental): Two eye drops containing PVP-Iodine instillation in the eye undergoing cataract surgery three times for three days before surgery.
  Each patient was evaluated for conjunctival flora variation by means of two conjunctival swabs before starting the treatment and at the end of the treatment before the surgery.
  Interventions: Device: IODIM

INTERVENTIONS:
Device: IODIM — Eye drops containing polyvinylpyrrolidone-Iodine (PVP-Iodine), hyaluronic acid and triglycerides

SUMMARY:
The purpose of the present study is to elucidate the qualitative and quantitative variation of ocular flora after treatment with eyedrops containing 0.6% povidone-iodine in the eye of patients undergoing routine cataract surgery.

DETAILED DESCRIPTION:
Two conjunctival swabs will be executed at 3 days before and at the day of routine cataract surgery in each eye of patients undergoing routine cataract surgery. After the collection of the first conjunctival swab a three-days treatment with eyedrops containing 0.6% povidone-iodine in the eye undergoing routine cataract surgery will be performed. Bacterial isolates will be identified by using standard microbiological protocols and total bacterial load will be determined at the two different time points. In vitro susceptibility testing to determine methicillin resistance in isolated Staphylococcus species will be performed. Controlateral eye of each patient will be used as control. Descriptive statistics will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Males and females aged between 40 and 80 years
* Patients who are candidates for cataract extraction

Exclusion Criteria:

* Males and females under 40 years and over 80 years
* Previous diseases of the eye, ocular surface and thyroid disease
* Known hypersensitivity to the product
* Presence of autoimmune diseases
* Pregnancy or breast-feeding
* Participation in other clinical studies

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
Variation of bacterial load of Positive Culture in Subjects Scheduled for Cataract Surgery | Three days of treatment
  Variation/Eradication of bacterial load in participants with positive culture at the screening visit. This variation/Eradication will be recorded at pre-surgical visit by means of a second collection of a conjunctival swab and culture analysis. This outcome will be assessed by comparing the number of participants undergoing eradication of their initial bacterial load or decrease of bacterial load after treatment.

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Oftalmologia Universitaria Ospedale Policlinico di Bari, Bari, BA
  - Ospedale Sacra Famiglia Fatebenefratelli, Erba, Como
  - Clinica Oculistica Azienda Ospedaliero-Universitaria, Presidio Ospedaliero G. Rodolico, Catania, CT
  - Centro di Microchirurgia Ambulatoriale di Monza, Monza, MB
  - Casa di Cura Villa Valeria di Roma, Roma, RM
  - Ospedale San Carlo di Nancy, Roma, RM